CLINICAL TRIAL: NCT05093244
Title: A Prospective, Randomized, Multi-center IDE Study to Assess the SeQuent Please ReX Drug Coated PTCA Balloon Catheter for the Treatment of In-stent Restenosis (RESPECT-ISR)
Brief Title: Resveratrol Excipient Paclitaxel Coated Balloon for Coronary Treatment
Acronym: RESPECT-ISR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to terminate study.
Sponsor: B. Braun Medical Inc. (Industry)
Collaborators: Bright Research Partners (Industry); Infraredx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIS-CL-5001
Record Dates: First submitted 2021-10-07; First posted 2021-10-26 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: In-stent Coronary Artery Restenosis; Coronary Artery Restenosis; In-stent Restenosis
Keywords: Drug coated balloon catheter; Paclitaxel coated balloon; Rapid exchange balloon tip catheter; Percutaneous transluminal coronary angioplasty; In-stent lesions in coronary arteries
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 2:1 ratio to either the SeQuent Please ReX or POBA arms, stratified by the presence or absence of baseline diabetes mellitus and acute coronary syndrome (ACS) vs. non-ACS presentation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SeQuent Please ReX (Experimental): Drug coated balloon (DCB) catheter.
  Interventions: Device: SeQuent Please ReX
- Plain old balloon angioplasty (POBA) (Active Comparator)
  Interventions: Device: Plain old balloon angioplasty (POBA)

INTERVENTIONS:
Device: SeQuent Please ReX — The SeQuent Please ReX is a conventional rapid exchange balloon tip catheter with a drug-coated balloon (DCB). The surface of the SeQuent Please ReX balloon is coated with paclitaxel, embedded in a soluble matrix (resveratrol).
  Arms: SeQuent Please ReX
Device: Plain old balloon angioplasty (POBA) — Any commercially available semi-compliant PTCA balloon may be used per the investigator's discretion.
  Arms: Plain old balloon angioplasty (POBA)

SUMMARY:
The objective of this study is to establish reasonable assurance of safety and effectiveness to support an FDA premarket approval (PMA) application for the SeQuent® Please ReX™ Drug Coated PTCA Balloon Catheter as indicated.

DETAILED DESCRIPTION:
The investigation is a prospective, randomized, multi-center IDE study comparing the SeQuent Please ReX to plain old balloon angioplasty (POBA). The study will be conducted at up to 30 investigational sites and enroll up to 296 patients with in-stent restenosis of a metallic coronary stent who are suitable candidates for PTCA procedures. After consent and assessment of inclusion and exclusion criteria, eligible patients will be randomized to either the SeQuent Please ReX or POBA arm based on a 2:1 randomization ratio. Subjects will return for follow-up through 5 years.

ELIGIBILITY:
INCLUSION CRITERIA:

1. ISR (>50%) of a metallic coronary stent of any type (BMS or DES)
2. Symptomatic ischemic heart disease, including:

   * Chronic stable angina (and/or objective evidence of myocardial ischemia on functional study or fractional flow reserve [FFR] measurement) or
   * Acute coronary syndrome (unstable angina or non-ST-elevation myocardial infarction (NSTEMI)), who require elective or urgent percutaneous coronary intervention (PCI)
3. One or two ISR lesions requiring treatment

   * ISR lesions may be located in two different vessels
   * Additional non-ISR (de novo) lesions are permitted and may be located in the target or other vessels
4. Target lesion reference vessel diameter is ≥2.0 or ≤4.0 mm by visual estimation
5. Total lesion length less than or equal to 34 mm by visual estimation (to permit treatment with balloon up to 40 mm)
6. Male or female, age 18 years or older
7. Willing to provide written informed consent and written HIPAA authorization prior to initiation of study procedures
8. Willing to comply with the specified follow-up visits
9. Willing and able to comply with post-treatment medications (dual antiplatelet therapy (DAPT) followed by life-long aspirin)
10. Non-target lesions must be treated successfully (i.e., residual diameter stenosis <30% without complications) before proceeding to treatment of ISR lesion(s)

EXCLUSION CRITERIA:

1. Target lesion has undergone more than two prior stent implant procedures, i.e., more than two layers of stent are present at any segment of target lesion
2. Presents with ST-elevation myocardial infarction (STEMI)
3. STEMI within the past 72 hours
4. Chronic kidney disease, defined as glomerular filtration rate (GFR) <15 ml/min/1.73m^2 on baseline labs
5. Thrombocytopenia, defined as a platelet count of <50,000 microL on baseline labs
6. Target lesion is a chronic total occlusion
7. Bleeding diathesis, coagulopathy, or contraindication to antiplatelet therapy
8. Target lesion restenosis is within a bio-resorbable scaffold
9. Target lesion is located within the left main
10. Pregnant (verified with a urine or blood pregnancy test), breast-feeding, or planning to become pregnant
11. Severely disabled and/or life expectancy appears limited (≤12 months) according to the investigator's opinion
12. Known hypersensitivity to paclitaxel and/or resveratrol or any of the product ingredients
13. Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints

Note: Bifurcation lesions are not excluded; however, the main branch should be treated per randomization, and the side branch should be treated provisionally per current standard of care.

Angiographic Exclusion Criteria:

Subjects must not meet any of the following angiographic exclusion criteria after lesion preparation:

1. Dissection type C - F
2. TIMI < III
3. Residual stenosis >30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Freedom from target lesion failure (TLF) | 12 months post-procedure
  TLF is defined as the composite of any of the following events:
  * Clinically-driven target lesion revascularization (TLR)
  * Myocardial infarction (MI; not clearly attributable to a nontarget vessel)
  * Cardiovascular death

SECONDARY OUTCOMES:
Late lumen loss (LLL) | 9 months post-procedure
  Assessed on the first 100 subjects reaching 9-month follow-up (angiographic cohort). Minimum lumen diameter (MLD) assessed at follow-up angiography minus the MLD assessed immediately after the index procedure. MLDs are measured by qualitative comparative analysis.
All death | 12 months post-procedure and annually thereafter to study completion
  Death of subject.
Cardiovascular death | 12 months post-procedure and annually thereafter to study completion
  Death resulting from cardiovascular causes.
Myocardial infarction (MI) | 12 months post-procedure and annually thereafter to study completion
  Not clearly attributable to a nontarget vessel
Major adverse cardiac events (MACE) | 12 months post-procedure and annually thereafter to study completion
  Defined as the composite of all death, clinically-driven TLR, and MI
Stent thrombosis | 12 months post-procedure and annually thereafter to study completion
  Early, late, or very late; ARC category of definite or probable
Clinically-driven target lesion revascularization (TLR) | 12 months post-procedure and annually thereafter to study completion
  Target lesion revascularization is defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Clinically-driven target vessel revascularization (TVR) | 12 months post-procedure and annually thereafter to study completion
  Target vessel revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion.
Device, lesion, and procedural success | Post-procedure (device and lesion success) and at discharge (procedural success)
  Device success defined as achievement of a final residual stenosis of ≤30% (as determined by the angiographic core lab), using the SeQuent Please ReX or control balloon. Lesion success defined as achievement of a final residual stenosis of ≤0% (as determined by the angiographic core lab), using any device. Procedural success defined as lesion success without the occurrence of major adverse events during the procedure, where "major adverse event" is considered to be an event without the occurrence of in-hospital MI, TVR, or cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Saucedo, MD, MBA, Principal Investigator — Froedtert & Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: No